CLINICAL TRIAL: NCT03956810
Title: Evaluation of the Prenatal Trip Assistance Pilot Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Erinn Hade, Associate Professor, New York University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2019H0009
Record Dates: First submitted 2019-05-15; First posted 2019-05-21 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Pregnancy Preterm; Infant Death
Keywords: transportation; prenatal care
MeSH Terms: conditions — Infant Death

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- On-demand transportation (Experimental): Women randomized to the intervention group will be able to contact the transportation broker via telephone, web portal, or the broker's mobile application. In addition to the current trips provided by their Medicaid managed care organization , women assigned to the intervention group will be provided with extra trips to the pharmacy and grocery store or food bank.
  Interventions: Other: On-demand transportation
- Usual transportation (Active Comparator): Women assigned to the usual care group will receive the usual transportation services from their Medicaid managed care organization.
  Interventions: Other: Usual transportation

INTERVENTIONS:
Other: On-demand transportation — On-demand scheduling via telephone, web portal, or the broker's mobile application.
  Arms: On-demand transportation
Other: Usual transportation — Usual transportation scheduling via call-center.
  Arms: Usual transportation

SUMMARY:
The prenatal trip assistance project is a study comparing two methods of delivering transportation assistance to pregnant women living in communities with high rates of infant mortality. Franklin County, Ohio, home of the state's capital of Columbus, has one of the highest rates of infant mortality in the U.S. at 8.2 per 1,000 live births.There have been many advances in "smart" applications in transportation over the past 10 years. However, despite the fact that the vast majority of impoverished women have a mobile phone, the transportation providers currently used by the Medicaid managed care plans are low tech with no mobile alerts or two-way communication with the woman. The purpose of the proposed study is to examine the preliminary efficacy of providing expanded and "smart" transportation services to increase communications, reliability, and customer satisfaction and reduce adverse pregnancy outcomes among women whose children are at high risk of infant mortality. The investigators aim to enroll and randomize 500 eligible pregnant women to either on-demand services or usual transportation services as provided by their Medicaid managed care organization. The primary outcome for the proposed trial will be overall satisfaction with transportation services as assessed by the final study questionnaire (i.e., two months after delivery or miscarriage) and secondary outcome measures will include: adequacy of prenatal care, preterm birth and infant mortality.

ELIGIBILITY:
Inclusion Criteria:

* Willing to consent to communication by phone, text, and email
* Access to a telephone (mobile or landline), tablet or computer
* Pregnant & <32 weeks of gestation
* Last menstrual period on or before 2/9/2020 or due by November 15, 2020
* At least 18 years old
* Enrolled in one of two Medicaid managed care organizations
* Residence in Franklin County, Ohio
* Ambulatory
* English speaking

Exclusion Criteria:

* No plans to move out of Franklin County prior to delivery
* Able to read, understand, and communicate in English
* Woman has not been previously enrolled in this study
* Race/ethnicity stratum is not full
* Willing to meet staff to be interviewed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
Satisfaction with transportation services: scale | Obtained 8 weeks postpartum
  Participants will be asked in one question to rate their level of overall satisfaction with transportation services measured on a five-point scale (5=very satisfied, 1=Very dissatisfied). Those who rate their satisfaction as either somewhat (4) or very satisfied (5) will be considered satisfied with transportation services in analysis.

SECONDARY OUTCOMES:
Kotelchuck Adequacy of Prenatal Care Utilization index | Through study completion, an average of 9 months after enrollment.
  The Adequacy of prenatal care utilization index, as defined by Kotelchuck (AJPH, 1994). This index utilizes information on: gestational age at entry to prenatal care, the number of prenatal care visits, and the gestational age at delivery (to determine an expected number of prenatal visits). The index includes two dimensions which are combined (adequacy of initiation of prenatal care and adequacy of received services) into a single summary prenatal care utilization index category (Adequate plus utilization, Adequate utilization, Intermediate utilization, Inadequate utilization).
The proportion of deliveries < 37 weeks gestation | Through study completion, an average of 9 months after enrollment.
  The proportion of preterm deliveries occurring before 37 weeks gestation
The proportion of infants who die within one year of birth | One year post delivery
  Death of a live born infant within the first year of life

CONTACTS AND LOCATIONS:
Overall Officials: Erinn M Hade, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No